CLINICAL TRIAL: NCT06019273
Title: Impacts of Different ART Regimens on Lipid Metabolism in People Living With Human Immunodeficiency Virus
Brief Title: Impacts of Different ART Regimens on Lipid Metabolism in People Living With HIV
Acronym: ART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: FAHZUIIT20220125B
Record Dates: First submitted 2023-08-16; First posted 2023-08-31 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: HIV Infection; Combined Antiretroviral Therapy
Keywords: HIV antiretroviral therapy lipid metabolism
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To compare the dynamic changes of lipid metabolism of people living HIV who treated with different antiretroviral therapy (ART) regimens such as Biktarvy EVG/c/TAF/FTC, DTG/FTC/TDF, TDF/3TC/EFV, etc. And to assess the safety and efficacy of different antiretroviral therapy.

DETAILED DESCRIPTION:
This was a prospective observational study aiming to evaluate dynamic changes of lipid metabolism in people living HIV who treated with different antiretroviral therapy (ART) regimens. At the same time, cardiovascular risk and the incidence of non-alcoholic fatty liver disease are assessed so as to compare the effects of different regimen on cardiovascular risk and NAFLD and hope to discover several cardiovascular risk-related individual lipid species.

ELIGIBILITY:
Inclusion Criteria:

1. People with HIV aged 18 years and older
2. Treated with stable antiretroviral therapy
3. Plasma HIV-1 RNA below 50 copies per milliliter for at least six months
4. Without other comorbidities or concomitant medications
5. Good compliance and can cooperated with the follow-up
6. Willing to participate in the study and sign informed consent.

Exclusion Criteria:

1. Pregnant or breast-feeding
2. Patients with poor treatment compliance
3. Patients refused to attend the regular follow-up examination
4. Patients with severe cardiovascular and cerebrovascular diseases or liver and kidney dysfunction
5. Acute infection (malaria, tuberculosis, helminthiasis, pneumonia, meningitis), moderate or severe malnutrition and diarrhea in the last 3 months
6. Take medications that may interfere with lipid metabolism throughout the study, such as statins/fibrates, antidiabetic
7. Participated in other clinical trials within 3 months.
8. Patients with severe mental illness

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients on stable antiretroviral therapy without any Acute infection or other complications. Any patient present meeting the inclusion criteria of the study will be offered to participate in the study.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2024-04-25 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Differences in lipid metabolism across ART treatment groups | 24 weeks, 48 weeks
  Morning fasting blood was drawn at the time of interview. lipidomic profile was identified by liquid chromatography-mass spectrometry (LC-MS). Change from baseline in lipidomic profile at 24 weeks and 48 weeks. Distinct lipidomic profile between different ART treatment groups at week 24 and week 48.

SECONDARY OUTCOMES:
conventional clinical lipid | 24weeks, 48weeks
  change from baseline in clinical blood lipid at 24 weeks and 48 weeks
levels of inflammatory cytokines | 24weeks, 48weeks
  The following inflammatory cytokines: interferon-alpha (IFN-α), TNF-α, IL-1, IL-6
T-cell subsets | 24weeks, 48weeks
  Absolute CD4+ and CD8+ T-cell counts and CD4/CD8 ratio were measured on peripheral blood mononuclear cells.
Immune activation | 24weeks, 48weeks
  Immune activation measured by the percentage of human leukocyte antigen-DR isotype (HLA-DR) and CD38 expressing T-cells in blood.
Gut microbiome | 24weeks, 48weeks
  Fecal samples of the participants were collected in sterile container before their clinic visits. The DNA was extracted using a QIAamp DNA stool mini kit. And gut microbiome was identified by using metagenome sequencing. Diversity and composition of gut microbiome in different groups at 24 weeks and 48 weeks
Tolerability and safety outcomes | 24weeks, 48weeks
  Discontinuation and occurrence of adverse event.
Cardiovascular Disease Risk | 24weeks, 48weeks
  the cardiovascular disease risk was determined by a Framingham cardiovascular risk score(FRS). Change from baseline in Framingham cardiovascular risk score at 24weeks and 48weeks The range of FRS is 0-100, participants are considered a higher 10-year cardiovascular risk who have a higher scores in FRS system
Nonalcoholic Fatty Liver Disease | 24weeks, 48weeks
  the nonalcoholic fatty liver disease was identified by hepatic steatosis index score.
  Change from baseline in incidence of Nonalcoholic fatty liver disease at 24weeks and 48weeks.
  The hepatic steatosis index (HSI) was used as a surrogate marker for non-alcoholic fatty liver disease (NAFLD). The range of HSI is 0-100. HSI = 8 × (ALT/AST) + BMI + (2, if diabetes mellitus) + (2, if female), with values < 30 ruling out and values>36 ruling in steatosis

CONTACTS AND LOCATIONS:
Locations (1):
- Zhikai Wan, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wan Z, Su J, Zhu X, Liu X, Guo Y, Xiang D, Zhou X, Peng X, Tao R, Cao Q, Lang G, Huang Y, Zhu B. Distinct Lipidomic Profiles between People Living with HIV Treated with E/C/F/TAF or B/F/TAF: An Open-Label Prospective Cohort Study. Infect Dis Ther. 2024 Apr;13(4):727-744. doi: 10.1007/s40121-024-00943-0. Epub 2024 Mar 15. PMID 38489119